CLINICAL TRIAL: NCT04505254
Title: Intermittent Therapy With the BTK Inhibitor Acalabrutinib (Calquence) in Combination With Obinutuzumab in Treatment Naive (Tn) Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Acalabrutinib and Obinutuzumab for the Treatment of Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1141; NCI-2020-05262 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1141 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-21; First posted 2020-08-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, obinutuzumab) (Experimental): Patients receive acalabrutinib PO BID every 12 hours starting on day 1 of cycle 1, and obinutuzumab IV over 4-6 hours on days 1 and 2 of cycle 3, and day 1 of cycles 4-8. Patients who do not achieve a complete response or remission after cycle 8 may receive single-agent acalabrutinib therapy PO BID for an additional 6 cycles at the discretion of their treating physician. Patients who are in partial response or who have stable disease receive an additional 6 cycles of acalabrutinib PO BID and obinutuzumab IV. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Biological: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759

SUMMARY:
This phase II trial investigates the how well acalabrutinib and obinutuzumab work in treating patients with chronic lymphocytic leukemia (CLL). Acalabrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with obinutuzumab may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving acalabrutinib and obinutuzumab may help to control disease progression in CLL patients who have not received treatment for CLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

• to determine the proportion of patients who have treatment-free remission 6 months after discontinuation of acalabrutinib plus obinutuzumab therapy.

SECONDARY OBJECTIVES:

* to determine clinical factors associated with a treatment-free remission of more than 6 months after discontinuation of acalabrutinib;
* to determine the treatment-free remission length;
* to evaluate the efficacy of re-treatment with acalabrutinib plus obinutuzumab in patients who experience disease relapse.

EXPLORATORY OBJECTIVES:

• to characterize the effects of limited duration acalabrutinib plus obinutuzumab therapy on the clonal architecture as determined by genome-wide genotyping and analysis (GWAs) and whole exome sequencing (WES) and to determine the frequency of BTK and PLCG2 mutation in patients relapsing after limited duration acalabrutinib plus obinutuzumab therapy.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice a day (BID) every 12 hours starting on day 1 of cycle 1, and obinutuzumab intravenously (IV) over 4-6 hours on days 1 and 2 of cycle 3, and day 1 of cycles 4-8. Patients who do not achieve a complete response or remission after cycle 8 may receive single-agent acalabrutinib therapy PO BID for an additional 6 cycles at the discretion of their treating physician. Patients who are in partial response or who have stable disease receive an additional 6 cycles of acalabrutinib PO BID and obinutuzumab IV. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis CLL/small lymphocytic lymphoma (SLL) and be untreated
* Patients must have an indication for treatment by 2018 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients of childbearing potential must be willing to practice highly effective birth control during treatment and for 2 days after the last dose of acalabrutinib or 18 months after the last dose of obinutuzumab, whichever is later
* A negative urine pregnancy test (within 7 days of day 1) is required for women with childbearing potential
* Adequate renal and hepatic function as indicated by all of the following: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) except for patients with bilirubin elevation due to Gilbert's disease who will be allowed to participate
* An alanine transferase (ALT) =< 2.5 x ULN
* An estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft-Gault equation unless disease related
* Free of prior malignancies for 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast who are eligible even if they are currently treated or have been treated and/or diagnosed in the past 2 years prior to study enrollment. If patients had another malignancy of indolent behavior in the past 2 years prior to study enrollment that is expected to be cured with treatment they received such patients can be enrolled, after consultation with the principal investigator

Exclusion Criteria:

* Pregnant or breast-feeding females
* Prior CLL/SLL treatment
* Known history of infection with human immunodeficiency virus (HIV) or any uncontrolled active significant infection (eg, bacterial, viral or fungal)
* Signs of active hepatitis B or C. Subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded
* Patients with uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP)
* Patients with severe hematopoietic insufficiency as defined by an absolute neutrophil count of less than 500/μL, unless disease-related, and/or a platelet count of less than 30,000/μL at time of screening for this protocol.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of heart failure, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation can enroll. Patients with a history of paroxysmal atrial fibrillation (PAF) or deep vein thrombosis or pulmonary embolism (DVT/PE) can be included if they had no signs of PAF or DVT/PE in the last 6 months before enrolment. Patients with ongoing atrial fibrillation (AFib) or ongoing PAF or DVT/PE should be excluded
* History of stroke or cerebral hemorrhage within 6 months
* Known history or evidence of bleeding diathesis or coagulopathy within 3 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 1. Bone marrow aspiration and/or biopsy are allowed
* Serious, non-healing wound, ulcer, or bone fracture
* Treatment with warfarin (Coumadin) or any other vitamin K antagonist. Patients who recently received warfarin must be off warfarin for at least 7 days prior to start of the study. Patients receiving novel oral anticoagulant (NOAC), also termed direct oral anticoagulant (DOAC) are permitted to enroll. Patients who are currently on a vitamin K antagonist must be switched to a non-vitamin K antagonist, such as a NOAC/DOAC
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components)
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) (in the absence of lupus anticoagulant) > 2 x ULN
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-free remission | At 6 months after discontinuation of acalabrutinib, up to 4 years
  Defined as the time from discontinuation of acalabrutinib to the date of CLL relapse with active disease.
Overall response rate | After 6 cycles (each cycle 28 days) of treatment,up to 4 years
  Defined as complete response
Overall response rate | After 6 cycles (each cycle 28 days) of treatment,up to 4 years
  Defined as partial response

SECONDARY OUTCOMES:
Clinical factors associated with a treatment-free remission | Up to 6 months after completion of treatment
  Will use Cox's proportional hazards analysis of predictors that have a p value < 0.2 in the univariate analysis. Explanatory variables that were highly correlated will be independently entered into the Cox's regression model. Factors significant in at least one model tested will be taken to be possible independent predictors of relapse risk. Demographic and clinical characteristics will be summarized using descriptive statistics, including means with standard deviations, or medians with ranges, histograms and box-plot. Fisher's exact test and Wilcoxon rank test will be used in the data analyses of categorical and continuous variables, respectively.
Treatment-free remission length | Up to 6 months after completion of treatment
  The median length of treatment-free remission will be estimated using the Kaplan-Meier method.
Success rate of re-treatment in patients who relapse | Up to 6 months after completion of treatment
  The success rate of re-treatment, along with the 95% confidence interval will be computed, and median length of treatment-free remission will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Burger, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org